CLINICAL TRIAL: NCT02381938
Title: Care2bWell: A Worksite Physical Activity & Wellness Program for Child Care Staff
Brief Title: Care2BWell: Worksite Wellness for Child Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-2438; 1R01HL119568 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-03-06 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Physical Activity
Keywords: inactivity; behavior change; worksite wellness; child care
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 6-month intervention to increase physical activity and improve other health related behaviors
  Interventions: Behavioral: Healthy Lifestyles
- Control (Other): 6-month intervention to educate and improve financial health
  Interventions: Other: Healthy Finances

INTERVENTIONS:
Behavioral: Healthy Lifestyles — 6-month intervention to increase physical activity and improve other health related behaviors
  Arms: Intervention
Other: Healthy Finances — 6-month intervention to educate and improve financial health
  Arms: Control

SUMMARY:
This study will evaluate the efficacy of a 6-month child care-based intervention to improve workers' physical activity and other health-related behaviors compared to an attention control intervention (Healthy Lifestyles vs. Healthy Finances). The study sample will use a cluster randomized design and a sample of 104 child care centers and 416 child care workers (4 workers/center). The intervention arm will receive a 6-month child care-based intervention designed to improve workers' moderate to vigorous physical activity (MVPA) and other health-related behaviors (Healthy Lifestyles). The control arm (attention control) will receive a similarly structured program about financial health (Healthy Finances). The primary outcome is workers' MVPA; and secondary outcomes include workers' dietary intake, weight, smoking, sleep, and stress, as well as the centers' health supportive policies/structures for staff wellness and the overall physical activity environment for children. All primary and secondary outcomes will be assessed at baseline, post-intervention (6 months), and maintenance (18 months).

DETAILED DESCRIPTION:
The proposed study will evaluate the efficacy of a 6-month, child care-based intervention to increase workers' MVPA and other health-related behaviors (Healthy Lifestyles) compared to an attention control condition (Healthy Finances). This study will use a two-arm, cluster-randomized controlled trial (RCT) and a sample of 104 child care centers and 416 workers (4 workers/center). The primary outcome will be workers' MVPA; and secondary outcomes include workers' weight, dietary intake, smoking status, sleep habits, and emotional health as well as child care centers' programs, policies and environment around worksite wellness and teachers' interactions with children around physical activity. All primary and secondary outcomes will be assessed at baseline, post-intervention (6 months), and maintenance (18 months).

For this study, 104 child care centers will be recruited from a mix of urban/suburban and rural areas. Potential child care centers in these counties will be identified using an online database of licensed child care facilities maintained by the North Carolina (NC) Division of Child Development and Early Education. State and local community partners will be engaged to help inform centers in targeted counties about the research study. Direct recruitment of centers will employ a variety of strategies (e.g., mail, email, telephone, website, video, in-person contacts). Once a center expresses interest, the center director will be engaged to recruit their staff (child care workers) to participate as a team.

Outcome Measures:

A series of measurements will be collected on participating child care center directors and staff at three time points - baseline, follow-up (6 months), and maintenance (18 months). Primary outcome measures will assess moderate to vigorous physical activity (MVPA) of center staff. Secondary outcomes measures will assess staff members' behavioral health risk factors as well as centers' programs, policies and environment around worksite wellness and teachers' interactions with children around physical activity. These measures will be collected during a one-day, on-site visit to the child care center, and supplemented with physical health assessments completed at the kick-off event. Center visits will be conducted by research assistants who have undergone extensive training and certification on all measurement procedures and are blinded to study-arm assignment. Similar data collection protocols will be used at all three time points - baseline, follow-up and maintenance.

Randomization:

Centers will be randomly assigned (1:1) into the intervention or control arm. Randomization will occur during local kick-off events (each center must attend one event). Each kick-off event will include a short wellness fair in the morning (including stations to collect baseline biomedical health assessments). Lunch will be provided, followed by random assignment into either the intervention or control arm. Timing allows for all of baseline measures to be complete prior to randomization. Centers in both the intervention and control arms will immediately start implementation of their respective programs.

Program Details/Intervention:

Healthy Lifestyles Intervention will kick off with an educational workshop and tailored feedback based on responses to the CHART assessment tool. The educational workshop and personalized health assessment summary will be delivered during the afternoon of the kick-off event in a group format with other participating centers. Following this launch, the intervention will provide 3 campaigns, each of which will include the following components: center support materials, director webinar, staff magazine, and behavioral goal setting/monitoring and weekly personalized feedback. The center support materials, director webinars, and staff magazines will be delivered directly to the center to support the center-based intervention. The behavioral goal setting/monitoring will be delivered directly to participating staff. While campaign structure is constant, topics of each campaign will vary. Campaign 1 focuses on increasing daily physical activity, cutting back on unhealthy snacking, and switching from sugary and diet drinks to water. Campaign 2 focuses on eating a diet rich in fruit and vegetables, whole grains, and lean protein, varying daily physical activity, and increasing strength training. Campaign 3 focuses on maintaining an active lifestyle, managing stress in a healthy way, and improving sleep habits.

Program Details/Control:

Healthy Finances Intervention will kick-off with an educational workshop and personalized health assessment snapshot at the kickoff community event. The educational workshop will be delivered during the afternoon of the kick-off event in a group format with other participating centers randomized to the Healthy Finances arm. The personalized health assessment snapshot will be provided during that workshop, but not reviewed in detail. It is intended to provide only a basic comparison of current behaviors to recommendations. Following this launch, the intervention will provide 3 campaigns, each of which will include the following components: director webinar, staff magazine, and a contest focused on quizzing knowledge gained from the magazines. The director webinars and staff magazines will be delivered directly to the center to support the center-based program. The contest and knowledge quizzes will be delivered directly to participating staff. While campaign structure is constant, topics of each campaign will vary. Campaign 1 focuses on the link between financial health and personal well-being (physical, mental), record-keeping: logging income and expenses, and thoughtful spending: creating and sticking to a spending plan. Campaign 2 focuses on creating and making the most of a personal savings account, and benefits of long-term investing: rules of thumb for picking investments. Campaign 3 focuses on understanding your credit report and credit score, understanding what good credit can do for you, and tips and strategies for improving your credit.

Analysis:

Investigators will compare the difference in mean change in MVPA between baseline and post intervention between Healthy Lifestyle and Healthy Finance arms, controlling for baseline physical activity. The primary analysis will test the hypothesis under the intent-to-treat principle using Generalized Linear Mixed Models (GLMM) that will account for the correlation induced by the clustering of staff within centers. Each GLMM will include a random intercept for centers (β 0) and fixed effects for the baseline value of the primary outcome (β1) and the intervention (β2) to test if the difference in mean change in the primary outcome is zero where β0 is the fixed intercept and e is error.

[Change in Primary Outcome6mo = β0 + β1PrimaryOutcomebaseline + β2Intervention + b0 + e] Including baseline score as a covariate in an analysis of covariance (ANCOVA), in our case a GLLM ANCOVA analysis, is a more powerful test than a group comparison of baseline to post-intervention change. Additionally, ANCOVA is not distorted by regression towards the mean bias, whereas a change analysis is. To further explore intervention effect, investigators will fit GLMMs that: 1) adjust for baseline covariates, considered a priori, to be relevant to change in MVPA; 2) adjust for baseline variables distributed differently between Healthy Lifestyle and Healthy Finance arms; 3) test interaction terms between treatment group and other covariates; and 4) examine completers only. While investigators will make every effort to minimize attrition at the center and participant level; some drop out is expected. Investigators will explore the potential bias from non-ignorable, non-response using two methods: 1) compare respondents and non- respondents to see if they differ systematically on values of non-missing variables; and 2) assess whether data are missing completely at random (MCAR), or missing at random (MAR) or missing not at random (MNAR) - non-ignorable. If missing data are ignorable (MAR and/or MCAR), investigators will consider imputing missing endpoint data using multiple imputation techniques. However, it is often hard to determine if missing data are ignorable; therefore, investigators will consider selection models (MNAR models) to assess if data are missing not at random and estimate the effect of the interventions after removing selection bias. Investigators will also consider using pattern mixture models to assess the sensitivity of our results to various assumptions of missing data patterns. Investigators' previous work in child care centers and worksites demonstrate good retention.

ELIGIBILITY:
Inclusion Criteria:

* Must have been in business for at least 2 years in order to demonstrate business stability and minimize participant loss-to-follow-up due to closing of centers.
* Must be planning to remain in business for at least the next 18 months to ensure our ability to collect follow-up data.
* Must have at least 4 workers (1 director/assistant director and 3 staff) who are willing to take part in the study and agree to study protocols - participation in three data collection time points, attendance at a kick-off event, and acceptance of random assignment.
* Center staff must speak and read English.

Exclusion Criteria:

* been in business for less than 2 years
* plans to close in the next 18 months
* director/assistant director unwilling to participate
* less than 3 child care staff willing to participate
* child care staff do not read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in moderate to vigorous physical activity (MVPA) | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Child care center staff members' MVPA will be assessed using accelerometers. Staff will wear a GT3X+ accelerometer for 7 days, for 24 hours a day (during all waking and sleeping hours), except when bathing or participating in swimming/water activities. Monitors will be programmed to sample acceleration at 30 Hz. Each monitor will be placed onto an adjustable belt that allows the monitor to be worn comfortably over the right hip. Adult cut-points will be applied to calculate minutes of sedentary, light, moderate and vigorous activity. Minutes of moderate to vigorous physical activity (MVPA) will be used as the primary outcome. Monitors will be distributed during the on-site visits to centers so that research assistants can adjust the belt to the appropriate length for each worker.

SECONDARY OUTCOMES:
Change in dietary intake | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Dietary intake will be assessed with a modified version of the Dietary Screener Questionnaire used in the National Health and Nutrition Examination Survey. Estimated intakes from this screener have moderate to high correlations (0.5 to 0.8) with estimated intakes from dietary recalls. The modified version used in this study will retain original items assessing fruits, vegetables, fiber/whole grains, added sugars, diary/calcium, and red and processed meat. In addition, some items will be merged (e.g., soda and sweetened fruit drinks asked as one item), others will be eliminated (e.g., salsa, pizza, tomato sauce), and a few new items will be added (e.g., dark green vegetables, eggs, lean meats, seafood, salty snacks, premade foods, dining out).
Change in smoking/e-cigarette status | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Use of tobacco and e-cigarettes will be assessed using four items, modified from the Behavioral Risk Factor Surveillance System Questionnaire. Items ask participants to estimate average use of tobacco and e-cigarettes based on their behavior during the past 30 days.
Change in sleep quality | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). Items ask participants to report on average hours of sleep per night and overall quality during the past month.
Change in stress | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Stress will be measured using items extracted from the Society for Behavioral Medicine's Common Data Elements, the Center for Epidemiologic Studies Depression Scale (CES-D), the Job Content Questionnaire, and previous studies. The CES-D is a assessment of depressive symptomology captures feeling of sadness, loss of interest, appetite disruption, sleep disruption, inability to think/concentrate, guilt, fatigue, agitation, and suicidal ideation. The Job Content Questionnaire assesses psychological demands resulting from one's job/occupation. For this study, items will be extracted to capture the constructs of psychological demands and decisional latitude.
Change in Body Mass Index | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Staff members' height and weight will be collected by trained research assistants during the center visit. Height will be measured to the nearest 1/8 inch with a Shorr measuring board (Shorr Productions, Olney, MD). Weight will be measured to the nearest 0.1 lb. with a Seca model 874 portable electronic scale (Seca Corporation, Columbia, MD). Height and weight measures will be used to calculate BMI (weight in kg/height in meters2) and weight status (underweight=BMI <18.5, normal weight = BMI 18.5-24.9, overweight = BMI 25.0-29.9, obese = BMI ≥30.0).
Change in waist circumference | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Staff members' waist circumference will be collected by trained research assistants during the center visit. Waist circumference will be measured to the nearest 0.1 cm with a Gulick II measuring tape.
Change in cardiovascular fitness | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Staff members' health will also be assessed with a series of biomedical health assessments which capture various indicators of fitness including cardiovascular fitness determined via resting/seated heart rate, resting/seated blood pressure and a 6-minute walk assessment. These assessments will be conducted by trained research assistants during the kick-off event.
Change in strength | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Staff members' health will also be assessed with a series of biomedical health assessments which capture various indicators of fitness including strength via the hand grip test. These assessments will be conducted by trained research assistants during the kick-off event.
Change in endurance | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Staff members' health will also be assessed with a series of biomedical health assessments which capture various indicators of fitness including endurance via the chair sit and stand test. These assessments will be conducted by trained research assistants during the kick-off event.
Change in balance | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Staff members' health will also be assessed with a series of biomedical health assessments which capture various indicators of fitness including balance via the 4-phase balance test. This assessment will be conducted by trained research assistants during the kick-off event.
Change in child care center worksite wellness environment | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Child care centers' programs, policies and environment around worksite wellness will be assessed with a Worksite Wellness Audit (WWA). The WWA has been developed specifically for this study, drawing on existing assessment protocols like the CDC Worksite Health Scorecard and Wisconsin's Worksite Assessment Checklist. The new tool will assess the five key elements which define a "comprehensive" wellness program (administrative supports, health education programs, environmental supports, linkage with other health programs, and screening + adequate follow-up). The WWA will incorporate three components: a director interview, an environmental scan, and a staff survey. Trained research assistants will conduct the director interview and environmental scan during the on-site visit. The staff survey will be completed as part of the online surveys.
Change in teacher physical activity practices | Measure collected 3-5 weeks prior to start of intervention and 1-5 weeks post intervention and repeated at 12-13 months post intervention
  Teachers' interactions with children around physical activity will be assessed using an extracted set of items from the Environment and Policy Assessment and Observation - Self-Report (EPAO-SR) protocol. These items will be presented as part of a paper survey, which trained research assistants will distribute to classroom teachers during the on-site visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dianne S Ward, EdD, Principal Investigator — University of North Carolina, Chapel Hill; Laura Linnan, ScD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Linnan LA, Vaughn AE, Smith FT, Westgate P, Hales D, Arandia G, Neshteruk C, Willis E, Ward DS. Results of caring and reaching for health (CARE): a cluster-randomized controlled trial assessing a worksite wellness intervention for child care staff. Int J Behav Nutr Phys Act. 2020 May 15;17(1):64. doi: 10.1186/s12966-020-00968-x. PMID 32414381